CLINICAL TRIAL: NCT05686837
Title: Prospective Healthcare-Associated Links in Transmission of Nontuberculous Mycobacteria Among People With Cystic Fibrosis
Brief Title: Prospective Healthcare-Associated Links in Transmission of Nontuberculous Mycobacteria
Acronym: pHALT NTM
Status: Enrolling by invitation | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Jewish Health (Other); University of Texas at Tyler (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-2792; HS-3175 (Other: BRANY)
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis; Nontuberculous Mycobacterial Pulmonary Infection
Keywords: epidemiology; outbreak investigation; transmission; acquisition; nontuberculous mycobacteria
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nontuberculous mycobacterial isolates from respiratory samples from people with CF will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People infected with NTM isolates identified in a cluster: All people with CF infected with NTM respiratory isolated identified in a cluster based on whole genome sequencing of the core genome will undergo epidemiologic investigation and home of residence watersheds will be mapped.
- People infected with NTM isolates not identified in a cluster: All people with CF infected with NTM respiratory isolated not identified in a cluster based on whole genome sequencing of the core genome will undergo epidemiologic investigation and home of residence watersheds will be mapped.

SUMMARY:
Pulmonary NTM infection is recognized as one of the most challenging infections to treat among people with cystic fibrosis (PwCF), notable for prolonged treatment courses and often poor response to therapy. Positive cultures for NTM occur in about 20% of children and adults with cystic fibrosis (CF). However, the source of NTM infection, modes of transmission, and exposure risks are poorly understood. It is thought that NTM is primarily acquired from environmental sites including soil and water as well as water supply systems to homes, hospitals, and clinics and from aerosols generated by flowing water from taps, showers, and fountains. Nonetheless, no direct molecular link has been established between environmental NTM and respiratory CF NTM. Healthcare-associated transmission of NTM among CF patients has been suspected and is of growing concern for CF Centers worldwide. Widespread global transmission of NTM, potentially via person-to-person transmission of fomites and aerosols has been reported. The parent HALT NTM study developed and published a standardized epidemiologic outbreak toolkit for investigation of healthcare-associated NTM outbreaks in CF Care Centers. The investigators are now moving to a prospective investigation, with the long-term goal of real-time early identification and mitigation of potential NTM outbreak investigations coupled with healthcare environmental sampling and home of residence watershed analysis of PwCF identified as belonging to an NTM cluster and receiving care at a single CF Care Center.

DETAILED DESCRIPTION:
This is a prospective, multicenter, nonrandomized study to investigate potential NTM outbreaks in the six CF Care Centers currently enrolled in the HALT NTM study. The study will investigate potential episodes of healthcare-associated NTM transmission and/or acquisition within participating U.S. Care Centers, coupled with healthcare environmental sampling and home of residence watershed analysis.

PART A / Epidemiologic Investigation:

The Colorado NTM Outcome Measure Advancement Core National Resource Centers (CO-NRC) provides a national reference laboratory for CF NTM. NTM respiratory isolates received from CF Care Centers around the U.S. undergo culture, molecular identification, antimicrobial susceptibility, and whole genome sequencing (WGS). Using this approach, the CO-NRC has identified clusters of NTM isolates, defined as highly similar strains at the genomic level, harbored by two or more people with CF (pwCF) who are cared for at the same CF Care Center. These identifications have heightened the concern for potential healthcare-associated NTM acquisition originating from patient-to- patient transmission or a common environmental source within Centers.

Using integrated clinical and epidemiological research methods, the parent HALT NTM study developed and validated a healthcare-associated epidemiologic investigation toolkit that can identify overlaps in source(s) of care between patients with highly similar NTM isolates in a Center. The parent HALT NTM toolkit facilitates a stepwise process by which individual Centers perform epidemiologic evaluation of patients identified by the CO-NRC as being infected with clustered NTM isolates.

The retrospective parent HALT NTM study of potential NTM outbreaks has been completed at six participating CF Care Centers. In the pHALT NTM study, participating sites will prospectively submit all respiratory NTM isolates from all PwCF receiving routine care over a two-year period to NJH Advanced Diagnostic Laboratories. All NTM isolates will be stored in the Biobank within the NTM Culture, Biorepository and Coordinating Core (Project ID: HS3149) and used for research purposes. The CO-NRC will utilize an honest broker to de-identify NTM isolates and will culture, bank, and extract DNA. The CO-NRC de-identified isolates will then be analyzed as previously described.

When highly related clusters are identified, the HALT NTM epidemiologic investigation toolkit will be independently used by each participating Center to identify overlaps in source(s) of care between patients with highly similar NTM isolates. Additionally, PwCF identified as being infected with highly similar NTM isolates will be asked to complete an online survey. The survey will ask the subject's basic demographic information, query their interactions with other PwCF, and document where they receive CF care.

PART B / Dust and Water Biofilm Collection:

Clustered NTM isolates could originate from a shared healthcare water source. Biofilms from healthcare dust and water supplies will be collected and NTM recovered, identified, and sequenced to determine if the respiratory CF NTM strain genotype is similar to those recovered from the healthcare dust and water supply.

Part C/Home of Residence Watershed Mapping: Clustered NTM isolates could originate from a shared home of residence water supply. PwCF having clustered NTM isolates will be asked to complete an online survey. The survey will ask subjects for their current and last 2 year's home address. The home of residence for PwCF identified in clusters will be extracted and geocoded to latitude and longitude coordinates and mapped to Hydrologic Unit Code level watersheds to determine if clustered PwCF share a common home of residence water supply source.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF consistent with the 2017 CFF guidelines.
* Male or female participant of any age who has a history of NTM or a first positive NTM culture collected as part of routine clinical care from expectorated sputum, induced sputum, throat/oropharyngeal swab and/or bronchoalveolar lavage.

Exclusion Criteria:

* No diagnosis of CF

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female participant of any age who has a history of respiratory NTM or a first positive NTM culture collected as part of routine clinical care from expectorated sputum, induced sputum, throat/oropharyngeal swab and/or bronchoalveolar lavage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic Investigation | 3 years
  Identification of a shared healthcare-associated source(s) between patients in a CF Care Center.
Dust and Water Biofilm Collection | 3 years
  Identification of healthcare dust and water biofilm NTM isolates that are highly related to the isolates recovered from PwCF.
Home of Residence Watershed Mapping | 3 years
  The primary endpoint is identification of common watersheds among pwCF infected with clustered NTM isolate.

SECONDARY OUTCOMES:
Epidemiologic Investigation | 3 years
  Incidence and prevalence of CF NTM species/subspecies by geographical region. Between Center comparisons of genetic similarity and patterns of potential transmission.
  Banking of isolates for ex vivo analysis.
Dust and Water Biofilm Collection | 3 years
  Incidence and prevalence of healthcare-associated dust and water biofilm NTM species/subspecies by geographical region.

CONTACTS AND LOCATIONS:
Overall Officials: Jane E. Gross, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (7):
- United States (7):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins Cystic Fibrosis Center, Baltimore, Maryland
  - Dell Children's Ascension, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Vermont Medical Center, Colchester, Vermont
  - UVA Health University Medical Center, Charlottesville, Virginia
  - UW Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All IPD will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will become available 9 months after publication and remain available for a total of 5 years.
Access Criteria: All IPD will be made available upon request. Deidentified individual data that supports the results will be shared beginning 9 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Result] Gross JE, Fullmer J, McClelland G, Caceres SM, Poch KR, Hasan NA, Jia F, Epperson LE, Lipner EM, Vang CK, Honda JR, Strand MJ, de Moura VCN, Daley CL, Strong M, Nick JA. Genomic and epidemiologic investigation of Mycobacterium abscessus isolates in a cystic fibrosis center to determine potential routes of transmission. J Cyst Fibros. 2025 Nov;24(6):1114-1123. doi: 10.1016/j.jcf.2025.07.003. Epub 2025 Aug 8. PMID 40783340
- [Result] Gross JE, Teneback CC, Sweet JG, Caceres SM, Poch KR, Hasan NA, Jia F, Epperson LE, Lipner EM, Vang CK, Honda JR, Strand MJ, Calado Nogueira de Moura V, Daley CL, Strong M, Davidson RM, Nick JA. Molecular Epidemiologic Investigation of Mycobacterium intracellulare Subspecies chimaera Lung Infections at an Adult Cystic Fibrosis Program. Ann Am Thorac Soc. 2023 May;20(5):677-686. doi: 10.1513/AnnalsATS.202209-779OC. PMID 36656594
- [Result] Gross JE, Caceres S, Poch K, Epperson LE, Hasan NA, Jia F, Calado Nogueira de Moura V, Strand M, Lipner EM, Honda JR, Strong M, Davidson RM, Daley CL, Nick JA. Prospective healthcare-associated links in transmission of nontuberculous mycobacteria among people with cystic fibrosis (pHALT NTM) study: Rationale and study design. PLoS One. 2023 Dec 20;18(12):e0291910. doi: 10.1371/journal.pone.0291910. eCollection 2023. PMID 38117792
- [Result] Gross JE, Finklea JD, Caceres SM, Poch KR, Hasan NA, Jia F, Epperson LE, Lipner EM, Vang CK, Honda JR, Strand MJ, Nogueira de Moura VC, Daley CL, Strong M, Nick JA. Genomic epidemiology of Mycobacterium abscessus at an adult cystic fibrosis programme reveals low potential for healthcare-associated transmission. ERJ Open Res. 2024 Jul 8;10(4):00165-2024. doi: 10.1183/23120541.00165-2024. eCollection 2024 Jul. PMID 38978544
- [Result] Gross JE, Caceres S, Poch K, Hasan NA, Davidson RM, Epperson LE, Lipner E, Vang C, Honda JR, Strand M, Strong M, Saiman L, Prevots DR, Olivier KN, Nick JA. Healthcare-associated links in transmission of nontuberculous mycobacteria among people with cystic fibrosis (HALT NTM) study: Rationale and study design. PLoS One. 2021 Dec 20;16(12):e0261628. doi: 10.1371/journal.pone.0261628. eCollection 2021. PMID 34929010
- [Result] Gross JE, Caceres S, Poch K, Hasan NA, Jia F, Epperson LE, Lipner E, Vang C, Honda JR, Strand M, Calado Nogueira de Moura V, Daley CL, Strong M, Davidson RM, Nick JA. Investigating Nontuberculous Mycobacteria Transmission at the Colorado Adult Cystic Fibrosis Program. Am J Respir Crit Care Med. 2022 May 1;205(9):1064-1074. doi: 10.1164/rccm.202108-1911OC. PMID 35085056